CLINICAL TRIAL: NCT06082999
Title: Gene-STEPS: Shortening Time of Evaluation in Paediatric Epilepsy Services: a Multi-centre Prospective Evaluation of the Impact of Early Genetic Diagnosis on Patient Outcomes
Brief Title: Gene-STEPS: Shortening Time of Evaluation in Paediatric Epilepsy Services
Acronym: Gene-STEPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Murdoch Childrens Research Institute (Other); The Hospital for Sick Children (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20NM24
Record Dates: First submitted 2023-08-31; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; Whole Genome Sequencing; Genetics; Paediatric
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA and RNA will be collected from patients. Blood samples for DNA will be collected from the parents of the patient, both in accordance with the patient consent form and information sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Overall, this observational cohort study aims too:

1. Implement rapid trio WGS for all children presenting to our health systems with epilepsy onset under 12 months of age.
2. Utilize electronic healthcare records and research databases to unite phenotypic and genomic data and to create a "virtual" registry across all institutions that will promote ongoing discovery.
3. Assess the impact of early genetic diagnosis on epilepsy, developmental, and health economic outcomes through formal longitudinal assessments of all children enrolled.

DETAILED DESCRIPTION:
In the past decade, the genomic revolution has led to the identification of underlying genetic aetiologies for childhood epilepsy, in the form of monogenic disorders affecting ion channels, neurotransmitter receptors, synaptic proteins, and other families of proteins. In a growing number of cases, the specific genetic diagnosis informs prognosis and genetic counselling, leads to the opportunity to participate in natural history studies, and even to changes in treatment that, to date anecdotally, may change outcomes in seizures and in neurodevelopment. However, a major challenge in clinical practice is that early intervention requires early diagnosis.

Currently the diagnostic odyssey in early-onset epilepsy is long and arduous for patients and their families. The timing and nature of genetic testing for such patients varies widely within and across countries and institutions. Our collective expertise includes epilepsy genetics research, genomic research, clinical epilepsy, clinical trials, and team science across four leading paediatric institutions in the IPCHiP Consortium: Boston Children's Hospital (US), Great Ormond Street Hospital and UCL Great Ormond Street Institute of Child Health (UK), Royal Children's Hospital Melbourne and Murdoch Children's Research Institute (Australia), and The Hospital for Sick Children ("Sick Kids", Canada). Each of our institutions has a proven track record of discovery and translation to patients, and our combined efforts in epilepsy will set a new standard for multi-institutional research, data sharing, and improvement. To investigate our hypothesis that rapid genetic diagnosis and tailored management could improve outcomes, we propose a novel approach to streamline and accelerate diagnostics in these severely affected children.

Overall, this observational cohort study aims too:

1. Implement rapid trio WGS for all children presenting to our health systems with epilepsy onset under 12 months of age.
2. Utilize electronic healthcare records and research databases to unite phenotypic and genomic data and to create a "virtual" registry across all institutions that will promote ongoing discovery.
3. Assess the impact of early genetic diagnosis on epilepsy, developmental, and health economic outcomes through formal longitudinal assessments of all children enrolled.

ELIGIBILITY:
Inclusion Criteria:

• Children under 12 months of age presenting with epilepsy.

Exclusion Criteria:

* Simple febrile seizures.
* Acute or remote symptomatic seizures due to sepsis, haemorrhage, cerebral infarction, hypoxic ischaemic encephalopathy or non-accidental injury.
* Structural malformations of the brain where the likely genetic cause is known such as tuberous sclerosis or lissencephaly.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with epilepsy onset under 12 months of age presenting to an epilepsy service. This is an international multi-centre collaborative study with GOSH as the UK sponsor.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of rapid genome sequencing in infantile epilepsy | Within three weeks of sample collection
  Feasibility is measured as the turnaround for participants, from both sample collection and seizure onset to GS result.
The Diagnostic Yield of rapid genome sequencing in infantile epilepsy | Within three weeks of sample collection
  The diagnostic yield is measured as the number of patients who receive a genetic diagnosis.
The immediate clinical utility of rapid genome sequencing in infantile epilepsy | Within one month of genetic result
  Clinical utility is measured as actual influence on treatment, potential for precision therapy, additional investigation indicated or avoided, additional prognostic information, influence on goals of care, or influence on genetic counselling (beyond recurrence risk). These are measured using The Clinician-reported Genetic testing Utility InDEx (C-GUIDE; Hayeems et al., 2022), as well as clinical data abstracted from health care records.

SECONDARY OUTCOMES:
The impact of early genetic diagnosis on developmental outcomes - Bayley 4 - Scales of Infant and Toddler Development. | At Recruitment, 12 and 30 months chronological age
  Bayley-4 items are scored 2 points for mastery of skill, 1 point for emerging skill and 0 points if skill is not present. Higher scores are, therefore, indicative of more advanced developmental abilities. Subtest standard scores range from 1 to 19, have a mean of 10 and a standard deviation of 3 (Bayley & Alyward, 2019).
The impact of early genetic diagnosis on developmental outcomes - Vineland Adaptive Behaviour Scales, Third Edition. | At Recruitment, 12 and 30 months chronological age
  The Vineland 3 generates five major domain composite scores: communication, daily living skills, socialisation, adaptive behaviour composite and motor skills, as well as a maladaptive score. Domain scores greater than or equal to 86 are considered adequate or above adequate. Domain scores less than or equal to 85 are considered moderately low-to-low, and indicate the patient has a significant skill deficit when compared with similarly aged peers. This is especially true for a domain score below 70. Maladaptive behavior scores up to 17 are considered average, scores of 18 to 20 are considered elevated and scores greater than 21 are considered clinically significant indicating a need for treatment intervention.
The impact of early genetic diagnosis on developmental outcomes - Gross Motor Function Classification System (GMFCS) | At Recruitment, 12 and 30 months chronological age
  The GMFCS is a standardised classification of functional motor abilities in children with cerebral palsy. Children are assigned a GMFCS level of 1-V according to motor functioning abilities. Level I represents the highest level of gross motor function and level V the lowest.
The impact of early genetic diagnosis on developmental outcomes - Paediatric Quality of Life Scale (PedsQL™) Infant Scales | At Recruitment, 12 and 30 months chronological age
  The PedsQL™ Infant Scales are a generic health related quality of life instrument specifically for healthy and ill infants ages 1-24 months. The PedsQL Infant Scales encompasses 5 scales: Physical functioning, physical symptoms, emotional functioning, social functioning and cognitive functioning. The Total Scale Score is computed as the sum of all items on the PedsQL™. Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL.
The impact of early genetic diagnosis on developmental outcomes - Parenting Stress Index, Fourth Edition Short Form | At Recruitment, 12 and 30 months chronological age
  The PSI-4 SF has thirty-six items are divided into three domains: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC), which combine to form a Total Stress scale. Percentile scoring: Between 16%-84% = Normal ranges of stress. Between 85%-89% = High levels of stress. Greater than or equal to 90% = Clinically significant.
The impact of early genetic diagnosis on epilepsy | 12 months and 30 months chronological age. The clinical dataset will also be retrieved at recruitment.
  Clinical Dataset & Seizure diary 4 weeks prior to visit
The views and experiences of parents offered rapid genomic sequencing for diagnosis of their child | For participating parents: 3-4 weeks and then 6 months after receiving GS result. For non-participating parents: 3 months after deciding not to participate.
  Qualitative interviews will be utilised to ascertain parents experiences of receiving the result, the impact of the result, and their hopes and concerns for the future. Parents who decline to participate will be asked about their decision not to take part in the study and have genome sequencing and suggestions for improving counselling and information.

CONTACTS AND LOCATIONS:
Overall Officials: Amy McTague, Principal Investigator — UCL Great Ormond Street Institute of Child Health
Locations (4):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Murdoch Childrens Research Institute, Parkville, Victoria, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- UCL Great Ormond Street Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided